CLINICAL TRIAL: NCT02352597
Title: Phytoestrogens as an Alternative to Estradiol in Reversing the Antiestrogenic Effect of Clomid on Endometrium in Ovulation Induction in Cases of Polycystic Ovarian Syndrome
Brief Title: Phytoestrogens as an Alternative to Estradiol in Ovulation Induction in PCOS
Acronym: PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 222
Record Dates: First submitted 2015-01-25; First posted 2015-02-02 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Polycystic Ovaries
Keywords: PCOS; Phytoestrogens; ovulation induction
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Phytoestrogens; Klimadynon; Estradiol; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- clomiphene citrate (Active Comparator): only50 mg orally every 8 hours started from cycle day 3 for 5 days
  Interventions: Drug: clomiphene citrate
- estradiol valerate and CC (Active Comparator): 2mg estradiol valerate orally daily from cycle day 7 - 11 in addition to CC
  Interventions: Drug: estradiol valerate; Drug: clomiphene citrate
- Phytoestrogen and CC (Active Comparator): 20mg of cimifuga racemosaorally from day 1- 12) in addition to CC
  Interventions: Drug: phytoestrogen; Drug: clomiphene citrate

INTERVENTIONS:
Drug: phytoestrogen — 20mg of cimifuga racemosa from day 1- 12
  Other Names: Klimadynon
  Arms: Phytoestrogen and CC
Drug: estradiol valerate — 2mg from cycle day 7 to day 11
  Other Names: cycloprogynova
  Arms: estradiol valerate and CC
Drug: clomiphene citrate — 50 mg orally every 8 hours started from cycle day 3 for 5 days
  Other Names: clomid

SUMMARY:
Prospective study conducted on 150 women with polycystic ovarian syndrome (PCOS) were randomly divided into 3 groups: group I (50 women) received clomiphene citrate (CC) only 50 mg orally every 8 hours started from cycle day 3 for 5 days, group II (50 women) received 2mg estradiol valerate daily from cycle day 7 - 11 in addition to CC and group III (50 women) received phytoestrogen (20mg of cimifuga racemosa from day 1- 12) in addition to CC.

DETAILED DESCRIPTION:
Prospective study conducted on 150 women with PCOS were randomly divided into 3 groups: group I (50 women) received CC only50 mg orally every 8 hours started from cycle day 3 for 5 days, group II (50 women) received 2mg estradiol valerate daily from cycle day 7 - 11 in addition to CC and group III (50 women) received phytoestrogen (20mg of cimifuga racemosa from day 1- 12) in addition to CC.

ELIGIBILITY:
Inclusion Criteria:

Women with both 1ry and 2ry infertility were included. All women were between 20 and 37 years old.

Exclusion Criteria:

women with endocrinological abnormalities as thyroid dysfunction or abnormal prolactin levels, those with hypothalamic or pituitary dysfunctions evaluated by low gonadotropin level, other causes of infertility as tubal factor evaluated by HSG or laparoscopy, abnormal uterine cavity evaluated by sonohystrography or hysteroscopy and male factor evaluated by semen analysis. Women with ovarian cysts were also excluded from the study

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
endometrial thickness | day 14 of menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school

IPD SHARING:
Plan to Share IPD: No